CLINICAL TRIAL: NCT00093899
Title: A Study to Evaluate the Efficacy and Safety of Ezetimibe/Simvastatin and Fenofibrate Coadministration in Patients With Mixed Hyperlipidemia
Brief Title: A Study to Evaluate an Investigational Drug in Patients With Mixed Hyperlipidemia (0653A-071)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0653A-071; 2004_044
Record Dates: First submitted 2004-10-07; First posted 2004-10-08 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hyperlipidemia; Hypercholesterolemia; Hypertriglyceridemia
Keywords: Mixed Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias; Hypercholesterolemia; Hypertriglyceridemia; Hyperlipoproteinemia Type II | interventions — Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: ezetimibe (+) simvastatin — Duration of Treatment: 6 months
  Other Names: MK0653A

SUMMARY:
The purpose of this study is to assess the cholesterol lowering effects of an investigational drug in patients with mixed hyperlipidemia (high cholesterol and high triglycerides).

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-79 years of age with high cholesterol and high triglycerides.

Exclusion Criteria:

* Individuals who do not meet specific cholesterol or triglyceride levels as required by the study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2004-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Plasma LDL-C.

SECONDARY OUTCOMES:
Plasma HDL-C, non-HDL-C, and TG. Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Farnier M, Roth E, Gil-Extremera B, Mendez GF, Macdonell G, Hamlin C, Perevozskaya I, Davies MJ, Kush D, Mitchel YB; Ezetimibe/Simvastatin + Fenofibrate Study Group. Efficacy and safety of the coadministration of ezetimibe/simvastatin with fenofibrate in patients with mixed hyperlipidemia. Am Heart J. 2007 Feb;153(2):335.e1-8. doi: 10.1016/j.ahj.2006.10.031. PMID 17239698
- [Background] Farnier M, Perevozskaya I, Taggart WV, Kush D, Mitchel YB. VAP II analysis of lipoprotein subclasses in mixed hyperlipidemic patients on treatment with ezetimibe/simvastatin and fenofibrate. J Lipid Res. 2008 Dec;49(12):2641-7. doi: 10.1194/jlr.P800034-JLR200. Epub 2008 Jul 31. PMID 18669979
- [Background] Gil-Extremera B, Mendez G, Zakson M, Meehan A, Shah A, Lin J, Mitchel Y. Efficacy and safety of ezetimibe/simvastatin co- administered with fenofibrate in mixed hyperlipidemic patients with metabolic syndrome. Metab Syndr Relat Disord. 2007 Dec;5(4):305-14. doi: 10.1089/met.2007.0011. PMID 18370800